CLINICAL TRIAL: NCT04952623
Title: Randomized Controlled Trial of Online Education for Physiotherapy Students to Improve the Management of Rotator Cuff Related Shoulder Pain
Brief Title: Online Education to Improve the Management of Rotator Cuff Related Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16.11.2020.95
Record Dates: First submitted 2021-06-17; First posted 2021-07-07 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2022-10

CONDITIONS: Subacromial Pain Syndrome; Rotator Cuff Injuries
Keywords: Online education; Shoulder pain; Physiotherapy
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-learning Group (Experimental): Participants will enroll in a 4-week e-learning program immediately after completing the pre-intervention assessment measures.
  Interventions: Other: Rotator Cuff Related Shoulder Pain E-Learning Program
- Wait-list Control Group (Active Comparator): Participants will enroll in a 4-week e-learning program, 4-5 weeks after completion of the pre-intervention assessment measures.
  Interventions: Other: Rotator Cuff Related Shoulder Pain E-Learning Program

INTERVENTIONS:
Other: Rotator Cuff Related Shoulder Pain E-Learning Program — The RCRSP e-learning program is designed according to the ADDIE Instructional Design Model in light of current literature.

SUMMARY:
A randomized controlled trial: Conservative treatments including physiotherapy and rehabilitation in the management of rotator cuff-related shoulder pain (RCRSP) are generally accepted as the first-line treatment approach, however, it is known that the disease-specific physiotherapy methods used by physiotherapists are highly variable. This may be caused by the insufficient knowledge of therapists about evidence-based interventions to RCRSP. The aim of this study is to develop the '' Rotator Cuff Related Shoulder Pain E-learning Program'' and evaluate its effect on students' knowledge and clinical reasoning skills related to evidence-based RCRSP interventions and their levels of confidence to have this knowledge compared with a control group.

DETAILED DESCRIPTION:
Shoulder pain is one of society's most common musculoskeletal problems, with a prevalence defined between 16-26%. Almost 70% of shoulder pain complaints are caused by pathologies associated with the rotator cuff. Conservative treatments including physiotherapy are widely accepted as a first-line treatment approach in the management of shoulder pain and on the other hand, the variety of physiotherapy practice is conspicuous. Despite the majority of physiotherapists provide treatment in line with current evidence, passive modalities are still highly preferred by some physiotherapists. The gap between research evidence and practice could be slightly due to the lack of an up-to-date undergraduate physiotherapy curriculum about the RCRSP. Therefore, the aim of this study is to develop the '' Rotator Cuff Related Shoulder Pain E-learning Program'' and evaluate its effect on students' knowledge and clinical reasoning skills related to evidence-based RCRSP interventions and their levels of confidence to have this knowledge compared with a control group. A randomized controlled trial including 146 4th grade physiotherapy students will be conducted. Students will be randomized into an e-learning group (n=73) or wait-list control group (n=73). The primary outcome will be the RCRSP achievement test, and the secondary outcome will be the self-reported confidence in knowledge and clinical reasoning skills related to RCRSP. All data will be collected through an online survey, which will be applied in two different time periods: pre-intervention and post-intervention. All groups will first answer the questionnaire at the beginning (week 0) and after the study group's e-learning activity (4-5 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 3th or 4th grade physiotherapy students

Exclusion Criteria:

* Students who are not currently enrolled in 3th or 4th grade

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Rotator cuff related shoulder pain achievement test | Change from baseline test scores at 4 weeks
  The RCRSP achievement test is consistent with 18 question items with multiple choices. The mean difficulty and KR-20 reliability coefficient of the test were calculated 0.59 and 0.84, respectively.

SECONDARY OUTCOMES:
Self-reported confidence in knowledge and clinical reasoning skills related to rotator cuff related shoulder pain | Change from baseline self-reported scores at 4 weeks
  The 3-item Questionnaire requires participants to rate their confidence in their knowledge and clinical skills related to RCRSP, using a 5-point Likert Scale ('not at all confident', 'not very confident', 'somewhat confident', 'confident' and 'very confident').

CONTACTS AND LOCATIONS:
Overall Officials: Mine Gülden Polat, PhD., Study Chair — Marmara University; Bahar Ayberk, PhD., Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No